CLINICAL TRIAL: NCT01770223
Title: An Open Label Study Assessing SVR and Viral Resistance Profile With Boceprevir Plus PEG-IFN Plus Ribavirin Triple Therapy in HCV-1 Infected Patients With Insulin Resistance Who Have Failed PEG-IFN Plus Ribavirin Dual Therapy
Brief Title: A Study of Viral Response to Triple Therapy in Hepatitis C Virus-Infected Participants With Insulin Resistance Who Failed Dual Therapy (MK-3034-113)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3034-113; 2012-002771-33 (EudraCT Number)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boceprevir + PegIFN-2b + RBV (Experimental): All participants will start treatment with 4 weeks of PegIFN-2b subcutaneously, 1.5μg/kg per week + RBV capsules orally, at a weight-based dose between 800-1400 mg/day divided into two daily doses (double therapy). Participants without cirrhosis will then continue on the PegIFN-2b and RBV with the addition of boceprevir capsules orally, 800 mg three times per day for 32 weeks (triple therapy), and will transition back to double therapy for the final 12 weeks of treatment (48 total weeks of therapy). Participants with cirrhosis or documented as null responders will receive triple therapy for 44 weeks (48 total weeks of therapy).
  Interventions: Drug: boceprevir; Biological: PegIFN-2b; Drug: RBV

INTERVENTIONS:
Drug: boceprevir
  Other Names: SCH 503034
Biological: PegIFN-2b
  Other Names: Peginterferon alfa-2b; PegIntron; SCH 054031
Drug: RBV
  Other Names: Ribavirin; Rebetol

SUMMARY:
This study is being done to find out if participants with insulin resistance and hepatitis C virus genotype 1 (HCV GT1) infections who failed dual therapy with peginterferon alfa (PegIFN) + ribavirin (RBV) will benefit from the addition of boceprevir to PegIFN + RBV (triple therapy).

ELIGIBILITY:
Inclusion criteria:

* Quantifiable serum hepatitis C virus-ribonucleic acid (HCV-RNA)
* Hepatitis C virus genotype 1
* Homeostasis Model of Assessment - Insulin Resistance (HOMA IR) > 2.5 in two determinations made 4 weeks apart (the first HOMA evaluation is able to be made 3 weeks before screening visit)
* Previous failure to achieve SVR with PegIFN plus ribavirin given for a minimum of 12 weeks without dose reduction below 80% of the adequate doses of the two drugs
* No response, partial response, or relapse after previous therapy
* Compensated liver disease with or without histologic or non-invasive evidence of liver cirrhosis
* If heterosexually active, a female participant of childbearing potential and a non-vasectomized male participant who has a female partner of childbearing potential must agree to use 2 effective contraceptives until 6 months after therapy has ended (7 months for male subject)

Exclusion criteria:

* Coinfection with HCV genotypes other than HCV-GT1
* Evidence of decompensated liver disease
* History of ascites, hepatic encephalopathy or of bleeding varices or severe portal hypertension
* History or signs or symptoms or evidence of hepatocellular carcinoma (HCC)
* History of organ transplant
* Coinfection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Severe psychiatric disease
* Inadequately controlled thyroid function
* Other important comorbidities (cardiovascular diseases, Type 1 diabetes or inadequately controlled type 2 diabetes, malignancies , etc)
* Substances abuse
* Alcohol intake >20 grams/day for females and >30 grams/day for males
* History of severe adverse events during previous treatment with PegIFN plus ribavirin including discontinuation of therapy for severe anemia or hematologic toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sustained virologic response (SVR) at 24 weeks after the end of 48 weeks of study treatment | Week 72

SECONDARY OUTCOMES:
Change from baseline in Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR) | Baseline up to 8 weeks